CLINICAL TRIAL: NCT00422500
Title: Longitudinal Study of the Prevalence, Severity, and Interference of Multiple Symptoms in Advanced Lung Cancer
Brief Title: Longitudinal Study of Multiple Symptoms in Advanced Lung Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2003-0701
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Advanced Lung Cancer; Chemotherapy Symptoms; Disease-Related Symptoms; Treatment-Related Symptoms; Symptom Management; Questionnaire; Telephone Interactive System; IVR Telephone System; DNA Repair Capacity; DRC; Cognitive Symptoms
MeSH Terms: conditions — Lung Neoplasms; Neurobehavioral Manifestations | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Study participants enrolled at M. D. Anderson will have additional serum drawn for cytokine analysis and DNA repair capacity. This blood will be drawn at the routine blood draws before treatment begins, and at the beginning of each treatment cycle.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chemotherapy Symptoms: Study participants with advanced-stage lung cancer.
  Interventions: Behavioral: Questionnaire; Behavioral: Telephone Interactive System; Other: Blood Samples

INTERVENTIONS:
Behavioral: Questionnaire — Surveys about symptoms, mood, and quality of life.
Behavioral: Telephone Interactive System — Automated telephone system call once a week during therapy, rating of severity of symptoms and daily life interference done with numeric key pad. Post therapy is complete, a call every two weeks for up to six months.
  Other Names: IVR Telephone System
Other: Blood Samples — For participating patients, 3 additional tablespoons of blood drawn at the beginning of each chemotherapy treatment (before treatment starts) and at the beginning of each cycle of treatment.

SUMMARY:
Primary Objectives:

* To compare the severity of symptoms, their impact on affective and health-related functional status, and symptom interference among patients with advanced-stage lung cancer following initiation of chemotherapy by disease status, tumor response to chemotherapy, and adequacy of symptom management.
* To examine the relationship of disease-related and treatment-related physical symptoms to affective impairment and the patient's reported symptom interference and functional impairment.
* To compare symptom severity, adequacy of symptom management, and interference with affective status and health-related function by patient's minority status.
* To explore the serum level of inflammatory cytokines during chemotherapy among lung cancer patients.
* To measure DNA repair capacity (DRC) in lymphocyte cultures of all patients enrolled in the protocol at baseline (before treatment) and during each follow-up blood draw. The hypothesis is that patients with suboptimal DRC will do better with chemotherapy than patients with efficient DRC.
* To extract DNA and genotype for polymorphisms in genes involved in the nucleotide excision repair pathway and in those involved in response to pain (opioid receptors, dopamine receptors, COMT). We hypothesize that:

  1. Polymorphisms in NER genes that modulate DNA repair capacity will also effect response to chemotherapy and to outcome.
  2. Cytokine gene polymorphisms account for variations in symptom outcomes (specific symptoms and symptom clusters) before, during and after chemotherapy.
  3. The COMT val/met polymorphism affects the metabolism of catecholamines on the modulation of response to sustained pain.
  4. Dopamine receptor polymorphisms that result in decreased density of dopamine receptors will result in a deficit in the dopamine pathway. that will also affect response to pain.
* To evaluate neurocognitive function to determine the prevalence, severity, and pattern of cognitive symptoms.

DETAILED DESCRIPTION:
One of the ways to learn about the symptoms of chemotherapy is by looking at how certain proteins called cytokines (found in the blood) change during therapy. Another way is to look at how symptoms change during treatment.

Before therapy starts, you will be asked to complete several questionnaires during a visit to the thoracic clinic at M. D. Anderson. These questionnaires measure physical and emotional (mental) symptoms. The questionnaires should take about 60 minutes to finish. You will also be asked to complete some cognitive (mental) questionnaires that take about 25 minutes to complete. During this visit, the research nurse will teach you how to use an interactive voice response telephone system for measuring symptoms. The research nurse will ask you the most convenient time for the telephone calls, and make sure the system is programmed to call you at that time. The date of the call will be at the same or close to the date of your weekly clinic visit.

Symptoms will be monitored weekly during chemotherapy treatment using this interactive voice response telephone system. The automated telephone system will call you once a week, and using the numeric key pad on your telephone, you will rate the severity of your symptoms and how much they interfere in your daily life. Once you complete therapy, the phone system will call every two weeks for up to six months. The information collected by these calls is only being used for this research study.

In addition to the telephone calls, the research nurse will arrange to meet you approximately every 6 weeks at your clinic visit. She will ask you to complete some surveys about your symptoms, mood, and quality of life. This meeting will take about 45 minutes. You will also be asked again to complete some cognitive (mental) questionnaires that take about 25 minutes to complete.

Research staff will also obtain from your medical record clinical information and lab values during your treatment period.

If you have agreed to participate in the companion caregiver study, the study staff will use your demographic and clinical data to study the influence of your symptoms on your caregiver's physical and mental health.

You are encouraged to report your symptoms to your treating physicians during the study, especially if you have any symptom that you rate greater than 7 on the 0 to 10 scale.

This is an investigational study. A total of up to 224 patients will take part in this multicenter study. Up to 112 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Is an adult > 18 years of age
2. Is diagnosed with Stage III or IV Lung cancer
3. Is scheduled for a new chemotherapy regimen. Patients who have received prior chemotherapy are eligible.
4. Is English- or Spanish-speaking
5. Currently lives in the United States

Exclusion Criteria:

1. Does not have access to telephones
2. Is unable to use the telephone interactive system
3. Has a current diagnosis of psychosis or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with advanced-stage lung cancer and disease- or treatment-related symptoms.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2003-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Longitudinal Data on Symptom Patterns + Severity | Total weekly IVR assessment period 18 weeks, generally include 6 cycles of chemotherapy and 2-3 assessments of response to chemotherapy.
  IVR telephone system to collect longitudinal data on symptom patterns and severity using patient tumor response evaluation after 2-3 cycles chemotherapy and total weekly IVR assessment period at 18 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Jackson Memorial Hospital, Miami, Florida
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org